CLINICAL TRIAL: NCT03126721
Title: A Phase 1, Open-label, Fixed-sequence Design Study To Assess The Effect Of Multiple Dose Administration Of Pf-06751979 On The Single Dose Pharmacokinetics Of Oral Midazolam In Healthy Adult Subjects
Brief Title: The Study is to Evaluate the Effect of Multiple Doses PF-06751979 on the Pharmacokinetics of Midazolam in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: B8271007; 2016-004238-50 (EudraCT Number)
Record Dates: First submitted 2017-04-14; First posted 2017-04-24 (Actual); Last update posted 2017-07-26 (Actual); Status verified 2017-07

CONDITIONS: Healthy
Keywords: drug interaction; PF-06751979; oral midazolam
MeSH Terms: interventions — Midazolam; PF-06751979

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- oral midazolam alone (Experimental): single dose of oral midazolam administered alone in period 1
  Interventions: Drug: midazolam
- oral midazolam administered with multiple doses of PF-06751979 (Experimental): single dose of midazolam on day 10 with multiple doses of PF-06751979 once a day on Days 1-11 in period 2
  Interventions: Drug: midazolam; Drug: PF-06751979

INTERVENTIONS:
Drug: midazolam — a single oral dose of 2 mg midazolam
Drug: PF-06751979 — multiple oral doses of PF-06751979 100 mg a day
  Arms: oral midazolam administered with multiple doses of PF-06751979

SUMMARY:
This is a drug interaction study to evaluate the PF-06751979 at steady state on the pharmacokinetics of oral midazolam single doses in fixed sequences including single dose midazolam alone in period 1 followed by multiple doses of 100 mg PF-06751979 once a day for 11 days with single dose midazolam co-administered on Day 10 in period 2

ELIGIBILITY:
Inclusion Criteria:

* Healthy female subjects of nonchildbearing potential and male subjects who, at the time of screening, are between the ages of 18 and 55 years, inclusive. Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure (BP) and pulse rate (PR) measurement, 12-lead electrocardiogram (ECG), or clinical laboratory tests.
* Body mass index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lb).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, (including alcoholic liver disease, nonalcoholic steatohepatitis (NASH), autoimmune hepatitis, and hereditary liver diseases), psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Any condition possibly affecting drug absorption (eg, gastrectomy).
* Treatment with an investigational drug within 30 days (or as determined by the local requirement) or 5 half-lives preceding the first dose of investigational product (whichever is longer).
* Subjects who have previously received PF-06751979.
* Fertile male subjects who are unwilling or unable to use a highly effective method of contraception as outlined in this protocol for the duration of the study and for at least 28 days after the last dose of investigational product.
* Use of prescription or nonprescription drugs and dietary supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of investigational product. As an exception, acetaminophen/paracetamol may be used at doses of <=1 g/day. Limited use of nonprescription medications that are not believed to affect subject safety or the overall results of the study may be permitted on a case-by-case basis following approval by the sponsor.
* Herbal supplements and hormone replacement therapy must have been discontinued at least 28 days prior to the first dose of investigational product.
* Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 60 days prior to dosing.
* History of hypersensitivity to midazolam or any other benzodiazapine.
* Other acute or chronic medical or psychiatric condition including recent (within the past year) or active suicidal ideation or behavior or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2017-04-18 (Actual); Primary Completion 2017-07-11 (Actual); Study Completion 2017-07-11 (Actual)

PRIMARY OUTCOMES:
midazolam Area Under the Curve from time 0 to last quantifiable concentration (AUClast) in Period 1 | 0, 0.5, 1, 2, 4, 6, 8, 10, 12, 16, 24 hrs post-dose
  the plasma midazolam AUC from 0 to tlast (time of last quantifiable concentration) when a single oral midazolam dose given alone
midazolam Cmax on Day 1 in Period 1 | 0, 0.5, 1, 2, 4, 6, 8, 10, 12, 16, 24 hrs post-dose
  the midazolam Cmax when single oral midazolam dose given alone
midazolam Area Under the Curve from time 0 to infinite (AUCinf) in Period 1 | 0, 0.5, 1, 2, 4, 6, 8, 10, 12, 16, 24 hrs post-dose
  the plasma midazolam AUC from 0 to infinity when a single oral midazolam dose given alone
midazolam AUClast in Period 2 | 0, 0.5, 1, 2, 4, 6, 8, 10, 12, 16, 24, 48 hrs post-dose
  the plasma midazolam AUC from 0 to tlast (time of the last quantifiable concentration) when a single oral midazolam given in presence of steady state PF-06751979
midazolam Cmax in Period 2 | 0, 0.5, 1, 2, 4, 6, 8, 10, 12, 16, 24, 48 hrs post-dose
  the midazolam Cmax when a single oral midazolam given in presence of steady state PF-06751979
midazolam AUCinf in Period 2 | 0, 0.5, 1, 2, 4, 6, 8, 10, 12, 16, 24, 48 hrs post-dose
  the plasma midazolam AUC from 0 to infinity when a single oral midazolam given in presence of steady state PF-06751979

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No
Information relating to our policy on data sharing and the process for requesting data can be found at the following link: http://www.pfizer.com/research/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B8271007&StudyName=A+Phase+1%2C+Open-label%2C+Fixed-sequence+Design+Study+To+Assess+The+Effect+Of+Multiple+Dose+Administration+Of+Pf-06751979+On+The+Single+Dose+Pharmacokinetics+Of+Oral+Midazolam+In+Healthy+Adult+Subjects